CLINICAL TRIAL: NCT06664333
Title: Experiences Reported by Siblings of Children Hospitalized in the PICU
Acronym: SIBCARE
Status: Recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Other Study IDs: APHP241201; 2024-A01918-39 (Other: ID RCB number)
Record Dates: First submitted 2024-10-28; First posted 2024-10-29 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-10

CONDITIONS: Intensive Care Pediatric
Keywords: Pediatric intensive care hospitalisation; Siblings; Semi-structured interviews; Post-traumatic stress disorder; Major depressive syndrome
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Siblings of pediatric intensive care hospitalized children: Siblings of children hospitalized in pediatric intensive care at Necker-Enfants Malades Hospital and Robert Debré Hospital, aged of 9 to 18 years old.
  Interventions: Other: Semi-structured interviews

INTERVENTIONS:
Other: Semi-structured interviews — The study consists of conducting two semi-structured interviews, with an estimated duration of 15 to 30 minutes, with siblings of children hospitalized in pediatric intensive care at Necker-Enfants Malades Hospital and Robert Debré Hospital.
  The first interview will take place during the stay in intensive care, the second 1 month after discharge from pediatric intensive care.

SUMMARY:
The care for a child in pediatric intensive care is recognized as a traumatic experience for the patient and their entourage. The needs and feelings of parents are relatively well supported in the literature. However, there is still too little data concerning siblings, who can nevertheless be impacted by this difficult life experience. The study consists of conducting two semi-structured interviews with siblings of children hospitalized in pediatric intensive care at Necker-Enfants Malades Hospital and Robert Debré Hospital. The first interview will take place during the stay in intensive care, the second one 1 month after discharge from pediatric intensive care.

DETAILED DESCRIPTION:
The care for a child in pediatric intensive care is recognized as a traumatic experience for the patient and their entourage. The needs and feelings of parents are relatively well supported in the literature. However, there is still too little data concerning siblings, who can nevertheless be impacted by this difficult life experience.

The study consists of conducting two semi-structured interviews, with an estimated duration of 15 to 30 minutes, with siblings of children hospitalized in pediatric intensive care at Necker-Enfants Malades Hospital and Robert Debré Hospital. The first interview will take place during the stay in intensive care, the second 1 month after discharge from pediatric intensive care.

The study will concern children and adolescents aged 9 to 18 years old because this is a population at risk in this situation. Concepts of illness, death and its irreversible nature evolve during childhood. By definition, there are three major stages which are: 0-6 years; 7-11 years; 10-18 years. For older children (> 10 years) these definitions are well established and they would be more at risk of presenting psychiatric disorders later (post-traumatic stress disorder, major depressive syndrome, etc.).

ELIGIBILITY:
Inclusion Criteria:

* Children and adolescents aged 9 to 18 years
* Whose sister or brother is hospitalized in pediatric intensive care at Necker-Enfants Malades hospital or Robert Debré hospital
* Holders of parental authority and children or adolescents informed and consenting to participate in the study

Exclusion Criteria:

* Death of patients
* Language barrier (French not mastered)
* Inability to participate in a semi-structured interview (intellectual disability)

Ages: 9 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children and adolescents aged 9 to 18 years whose sister or brother is hospitalized in pediatric intensive care at Necker-Enfants Malades hospital or Robert Debré hospital.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2025-01-21 (Actual); Primary Completion 2027-12-21 (Estimated); Study Completion 2027-12-21 (Estimated)

PRIMARY OUTCOMES:
Needs reported by children | 1 month
  Qualitative interpretation of the responses given by children during the two interviews.

SECONDARY OUTCOMES:
Assessment of the impact on the daily life of siblings following their visit to the intensive care unit | 1 month
  Assessment of the impact on the daily life of siblings following their visit to the intensive care unit to see their brother/sister.
  Qualitative interpretation of the responses given by children during the two interviews.
Assessment of the feelings during the visit of children and adolescents following the hospitalization of their brother or sister in pediatric intensive care | 1 month
  Assessment of the feelings during the visit of children and adolescents following the hospitalization of their brother or sister in pediatric intensive care.
  Qualitative interpretation of the responses given by children during the two interviews.
Assessment of the medium-term impact on the daily life of siblings after the discharge of their brother or sister from intensive care | 1 month
  Assessment of the medium-term impact on the daily life of siblings after the discharge of their brother or sister from intensive care.
  Qualitative interpretation of the responses given by children during the two interviews.

CONTACTS AND LOCATIONS:
Overall Officials: Léo MD Berger, Doctor, Principal Investigator — Assistance Publique - Hôpitaux de Paris; Agathe MD Béranger, Doctor, Study Director — Assistance Publique - Hôpitaux de Paris
Locations (2):
- France (2):
  - Hôpital Necker-Enfants Malades, Paris
  - Hôpital Robert Debré, Paris

REFERENCES:
- [Background] Youngblut JM, Brooten D. What Children Wished They Had/Had Not Done and Their Coping in the First Thirteen Months after Their Sibling's Neonatal/Pediatric Intensive Care Unit/Emergency Department Death. J Palliat Med. 2021 Feb;24(2):226-232. doi: 10.1089/jpm.2019.0538. Epub 2020 Jul 8. PMID 32640860
- [Background] Brooten DA, Youngblut JM, Roche RM, Caicedo CL, Page TF. Surviving Siblings' Illnesses, Treatments/Health Services over 13 Months after a Sibling's Death. J Child Fam Stud. 2018 Jun;27(6):2049-2056. doi: 10.1007/s10826-018-1044-1. Epub 2018 Mar 19. PMID 30766016
- [Background] Lovgren M, Jalmsell L, Eilegard Wallin A, Steineck G, Kreicbergs U. Siblings' experiences of their brother's or sister's cancer death: a nationwide follow-up 2-9 years later. Psychooncology. 2016 Apr;25(4):435-40. doi: 10.1002/pon.3941. Epub 2015 Aug 11. PMID 26260031
- [Background] Abela KM, Wardell D, Rozmus C, LoBiondo-Wood G. Impact of Pediatric Critical Illness and Injury on Families: An Updated Systematic Review. J Pediatr Nurs. 2020 Mar-Apr;51:21-31. doi: 10.1016/j.pedn.2019.10.013. Epub 2019 Dec 23. PMID 31874458
- [Background] Abela KM, Casarez RL, Kaplow J, LoBiondo-Wood G. Siblings' experience during pediatric intensive care hospitalization. J Pediatr Nurs. 2022 May-Jun;64:111-118. doi: 10.1016/j.pedn.2022.02.008. Epub 2022 Mar 11. PMID 35287059
- [Background] Gonzalez-Dambrauskas S, Mislej C, Vasquez-Hoyos P, Rotta AT. Family Presence and Visitation Practices in Latin American PICUs: An International Survey. J Pediatr Intensive Care. 2020 Sep 14;10(4):276-281. doi: 10.1055/s-0040-1716831. eCollection 2021 Nov. PMID 34745701
- [Background] Davidson JE, Aslakson RA, Long AC, Puntillo KA, Kross EK, Hart J, Cox CE, Wunsch H, Wickline MA, Nunnally ME, Netzer G, Kentish-Barnes N, Sprung CL, Hartog CS, Coombs M, Gerritsen RT, Hopkins RO, Franck LS, Skrobik Y, Kon AA, Scruth EA, Harvey MA, Lewis-Newby M, White DB, Swoboda SM, Cooke CR, Levy MM, Azoulay E, Curtis JR. Guidelines for Family-Centered Care in the Neonatal, Pediatric, and Adult ICU. Crit Care Med. 2017 Jan;45(1):103-128. doi: 10.1097/CCM.0000000000002169. PMID 27984278
- [Background] McPeake J, Castro P, Kentish-Barnes N, Cuzco C, Azoulay E, MacTavish P, Quasim T, Puxty K. Post-hospital recovery trajectories of family members of critically ill COVID-19 survivors: an international qualitative investigation. Intensive Care Med. 2023 Oct;49(10):1203-1211. doi: 10.1007/s00134-023-07202-9. Epub 2023 Sep 12. PMID 37698596
- [Background] Kentish-Barnes N, Cohen-Solal Z, Morin L, Souppart V, Pochard F, Azoulay E. Lived Experiences of Family Members of Patients With Severe COVID-19 Who Died in Intensive Care Units in France. JAMA Netw Open. 2021 Jun 1;4(6):e2113355. doi: 10.1001/jamanetworkopen.2021.13355. PMID 34152418
- See also: Ricignuolo C, Fostini O. Quelle place pour les frères et sœurs ?: Histoire de la première rencontre entre la fratrie et le nouveau-né hospitalisé. Carnet PSY [Internet]. 1 nov 2013 [cité 2 juill 2024];N° 175(8):35-7 — https://shs.cairn.info/revue-le-carnet-psy-2013-8-page-35?lang=fr&ref=doi